CLINICAL TRIAL: NCT00678483
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter, Multinational Study to Assess the Long-Term Effect, Over 1 Year, of Rimonabant 10 mg in Comparison With Rimonabant 20 mg After an Initial Treatment Period of 6 Months With Rimonabant 20 mg in Overweight or Obese Patients
Brief Title: Long-Term Effect of 10 mg Versus 20 mg Rimonabant in Overweight or Obese Patients
Acronym: MODERATO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: ICD, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10139; EudraCT : 2007-002492-14
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Obesity; Weight Loss
Keywords: Cholesterol; HDL; triglycerides; insulin; blood glucose
MeSH Terms: conditions — Obesity; Weight Loss; Insulin Resistance | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 10 mg
  Interventions: Drug: rimonabant (SR141716)
- 2 (Experimental): 20 mg
  Interventions: Drug: rimonabant (SR141716)

INTERVENTIONS:
Drug: rimonabant (SR141716) — once daily

SUMMARY:
The primary objective of this study is to assess, over a period of 12 months, the effect on weight loss and weight maintenance of rimonabant 10 mg in comparison with rimonabant 20 mg in overweight/obese patients after an initial treatment period of 6 months with rimonabant 20 mg.

Secondary objectives are to assess the effect of rimonabant over a period of 12 months on waist circumference, high-density lipoprotein (HDL)-Cholesterol and triglycerides (TG), fasting plasma glucose (FPG), fasting insulin and to evaluate the long-term safety and tolerability of rimonabant 10 mg and 20 mg over a period of 12 months after randomization in overweight/obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index (BMI) of at least 30 kg/m² or BMI >27 kg/m² with associated risk factors such as type 2 diabetes or dyslipidemia

Exclusion Criteria:

* Weight loss > 5 kg within 3 months prior to screening Visit.
* Presence of any clinically significant endocrine disease including the presence of type 1 diabetes
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safe participation including uncontrolled serious psychiatric illness such a major depression within the last 2 years, and history of other severe psychiatric disorders
* Previous participation in a clinical study with rimonabant
* Administration of other investigational drugs, anti-obesity drugs or other drugs for weight reduction
* Pregnancy and absence of effective contraceptive method for females of childbearing potential
* Exenatide
* Insulin therapy
* Recent change or need for change in the oral antidiabetic treatment
* Recent change or need for change in the lipid lowering treatment
* Presence of severe renal or hepatic impairment

The above information is not intented to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in weight from baseline to 12 months | 12 months

SECONDARY OUTCOMES:
Efficacy: - Absolute change in waist circumference from baseline - Relative change in HDL-Cholesterol and in Triglycerides from baseline - Absolute change in Fasting Plasma Glucose from baseline | 12 months
Safety : Vital signs, adverse events, laboratory tests | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi- Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Bucharest, Romania